CLINICAL TRIAL: NCT01457274
Title: A Randomised Controlled Trial of "Light" Versus "Deep" Sedation for Elective Outpatient Colonoscopy: Recall, Procedural Conditions and Recovery
Brief Title: "Light" Versus "Deep" Bispectral Index (BIS) Guided Sedation for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Principal Investigator, Associate Professor Kate Leslie, Head of Reaseach and Staff anaesthetist, The Royal Melbourne Hospital, Melbourne Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2011.066
Record Dates: First submitted 2011-09-22; First posted 2011-10-21 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Anaesthesia
Keywords: AMBULATORY CARE; AWARENESS AND RECALL; Propofol; Patient Safety and Satisfaction; Colonoscopy; Elective outpatient colonoscopy; Procedural sedation
MeSH Terms: conditions — Personal Satisfaction | interventions — Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- "light" sedation (Experimental): In this study the depth of sedation will be guided by the Bispectral Index monitor (BIS monitor). A BIS value of 70-80 will be targeted in the "light" sedation arm.
  Interventions: Other: Sedation depth
- "deep" sedation (Active Comparator): In this study the "deep" sedation arm will have a BIS value of less than 60 targeted.
  Interventions: Other: Sedation depth

INTERVENTIONS:
Other: Sedation depth — The intervention is the depth of sedation targeted in this study.
  Patients enrolled in this study will be sedated with the same medications (fentanyl bolus and propofol target controlled infusion), and at the same starting doses, in each study arm. However, the depth of sedation targeted will differ between the arms, and this depth will be guided by the BIS monitor.
  It is expected that those patients randomised to "deep" sedation will require a higher dose of sedative medication to achieve their target BIS value (<60) than those in the "light" sedation group (BIS 70-80).
  Other Names: BIS monitor; Bispectral index; Aspect medical

SUMMARY:
In this trial, patients undergoing elective colonoscopy under sedation will be randomised to BIS-guided sedation targeting either "light" (bispectral index [BIS] 70-80) or "deep" (BIS<60) sedation. Sedation will be achieved with a standardised regimen of target-controlled infusion of propofol and fentanyl bolus. The primary end point will be the incidence of procedure recall in each group - this will be assessed at the conclusion of the procedure. The procedural conditions, cardio-respiratory complications and recovery including cognitive function will be assessed during and immediately after the procedure. The incidence of dreaming and patient satisfaction with anaesthesia care will be recorded immediately after the procedure. The study will be complete when the patient leaves the hospital on the day of the procedure.

DETAILED DESCRIPTION:
Controversy exists about the need for deep sedation or light sedation during elective colonoscopy. Deep sedation ensures amnesia for the procedure and may ensure better operating conditions, but may result in cardiorespiratory side effects and prolonged recovery. Differences exist between countries regarding the prevailing depth of sedation with deeper sedation in general being administered in Australia than the United States. This study aims to explore that controversy.

ELIGIBILITY:
Inclusion Criteria:

* Plan for elective outpatient colonoscopy under sedation
* Able and willing to provide written informed consent for study entry and completion of all study related procedures
* American Society of Anesthesiologists' (ASA) physical status grade 1-3

Exclusion Criteria:

* Colonoscopy and gastroscopy booked as joint procedures
* Colonoscopy on emergency patients and/or inpatients
* Inadequate English comprehension (verbal and written to understand the Participant Information and Consent Form)
* Intellectual or psychiatric disability that prevents consent to and comprehension of study procedures
* Significant cognitive impairment that prevents independent conduct of activities of daily living or results in 3rd party procedural consent being obtained
* ASA physical status grade 4-5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Recall of procedure | 1 day. Day of procedure
  Upon rousing patients will be asked if they remember anything between the commencement of sedation and when they awoke from sedation

SECONDARY OUTCOMES:
Complications | 1 day. Day of procedure only.
  The treating anaesthetist will record if any of the following complications occur during the sedation for colonoscopy.
  1. Hypoxia
  2. Airway obstruction
  3. Hypotension
  4. Bradycardia
  5. Agitation
Speed and quality of recovery | 1 day. Day of procedure only. Measured before discharge from hospital
  Time from starting sedation until opening eyes in the post anaesthesia care unit, and time until readiness for hospital discharge will be recorded.
  Cognitive function at hospital discharge, compared to pre-procedure function, will be assessed by the CogState(TM) test battery.
Satisfaction | 1 day. Day of procedure only. Measured before discharge from hospital
  Proceduralist and anaesthetist satisfaction with the sedation will be recorded at the end of the procedure.
  Patient satisfaction with their anaesthesia care will be assessed at the time they are ready for hospital discharge.
Dreaming | 1 day. Day of procedure.
  Upon rousing in the post anaesthesia care unit patients will be asked the modified Brice questionnaire ("What is the last thing you remember before you went to sleep?", "What is the first thing you remember when you woke up?", "Did you remember anything in between?", and "Did you have any dreams?").
  Dreaming will be assessed by the response to quesion 4.

CONTACTS AND LOCATIONS:
Overall Officials: Megan L Allen, BMBS, Principal Investigator — Melbourne Health; Kate Leslie, MBBS, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne Hospital, Parkville, Victoria, Australia